CLINICAL TRIAL: NCT00054132
Title: A Phase II Study of OSI-774 in Combination With Bevacizumab in Patients With Stage IV Breast Cancer
Brief Title: Erlotinib Hydrochloride and Bevacizumab in Treating Patients With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-02225; NCI-2013-02225 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000269900; 02-119; MSKCC-02119; NCI-5761; 02-119 (Other: Memorial Sloan-Kettering Cancer Center); 5761 (Other: CTEP); N01CM17105 (NIH); P30CA008748 (NIH)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Recurrent Breast Carcinoma; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (erlotinib hydrochloride, bevacizumab) (Experimental): Patients receive erlotinib hydrochloride PO QD on days 1-21 and bevacizumab IV over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Bevacizumab; Drug: Erlotinib Hydrochloride; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF rhuMAb; Avastin; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF
Drug: Erlotinib Hydrochloride — Given PO
  Other Names: Cp-358,774; OSI-774; Tarceva
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies how well erlotinib hydrochloride and bevacizumab work in treating patients with stage IV breast cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as bevacizumab, may interfere with the ability of tumor cells to grow and spread. Giving erlotinib hydrochloride and bevacizumab may be an effective treatment for breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of bevacizumab in combination with OSI-774 (erlotinib hydrochloride) in patients with previously treated metastatic breast cancer, as measured by objective response rate.

SECONDARY OBJECTIVES:

I. To determine the toxicity of bevacizumab in combination with OSI-774 in patients with previously treated metastatic breast cancer.

II. To evaluate the efficacy of bevacizumab in combination with OSI-774 in patients with previously treated metastatic breast cancer, as measured by time to disease progression, duration of response and the proportion of patients with stabilization of disease >= 6 months.

III. To determine the molecular profile of the patient's primary breast tumor, and to explore the relationship between these molecular characteristics and the response to treatment.

IV. To explore changes in biological markers in pre- and post-treatment tumor tissue in a subset of patients with accessible sites of disease.

V. To explore a pre- and post-treatment analysis of circulating endothelial cells and the relationship of this analysis to serum markers of angiogenesis as well as response to treatment.

VI. To obtain serial measurements of circulating epithelial cells and explore the relationship of these cells with circulating endothelial cells, markers of angiogenesis, and epidermal growth factor receptor (EGFR) expression.

OUTLINE:

Patients receive erlotinib hydrochloride orally (PO) once daily (QD) on days 1-21 and bevacizumab intravenously (IV) over 30-90 minutes on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed carcinoma of the breast with metastatic (stage IV) disease that is currently stable or progressing after therapy
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques or as >= 10 mm with spiral computed tomography (CT) scan
* Patients must have either stable disease or disease progression on or after therapy with one or two conventional chemotherapy regimens for the treatment of metastatic (stage IV) breast cancer

  * Prior treatment with high-dose chemotherapy and autologous stem cell/bone marrow transplantation is allowed, and is considered one prior regimen when administered for metastatic disease
  * There is no restriction for the number of prior hormonal therapies or immunotherapies
  * If human epidermal growth factor receptor 2 (Her2)/neu-positive (defined as 3+ by immunohistochemistry [IHC] or positive by fluorescence in situ hybridization [FISH]), prior therapy with trastuzumab required
  * Any number of prior regimens of chemotherapy and/or hormonal therapy are allowed in the adjuvant setting, and do not count towards prior therapy when determining eligibility for this trial
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Life expectancy of greater than 3 months
* Leukocytes >= 3,000/ul
* Absolute neutrophil count >= 1,000/ul
* Platelets >= 75,000/ul
* Total bilirubin within normal institutional limits
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT[) =< 2.5 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min for patients with creatinine levels outside institutional normal using the Cockcroft-Gault formula
* Women of childbearing potential must agree to use adequate contraception (barrier method of birth control) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must have breast cancer tissue available as either paraffin blocks or unstained slides for planned correlative science sub study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, radiotherapy immunotherapy or investigational therapy within 3 weeks prior to starting treatment (6 weeks for nitrosoureas or mitomycin C), or hormonal therapy within 2 weeks prior to starting treatment
* Patients may not be receiving any other investigational agents
* History or evidence upon physical examination of central nervous system (CNS) disease (e.g., primary brain tumor, seizures not controlled with standard medical therapy, any brain metastases, or history of stroke); all subjects must have a baseline CT or magnetic resonance imaging (MRI) of the head
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to OSI-774 or bevacizumab
* Prior treatment with kinase insert domain receptor (KDR) inhibitors (e.g. vascular endothelial growth factor [VEGF] Trap, Su5416, Su6668, ZD6474, PTK757, IMC-1CII)
* Prior treatment with EGFR targeting therapies (e.g. ZD1839 or C225)
* Major surgery, open biopsy or significant traumatic injury occurring within 28 days prior to treatment; this does not apply to indwelling catheters, which require an interval of at least 24 hours between placement of the catheter and treatment with bevacizumab
* Current or recent (within 10 days prior to treatment) use of full-dose oral or parenteral anticoagulants or thrombolytic agents (except as required to maintain patency of preexisting, permanent indwelling IV catheters; for subjects receiving warfarin, international normalized ratio [INR] should be < 1.5)
* Chronic daily treatment with aspirin (> 325 mg/day) or nonsteroidal anti-inflammatory medications known to inhibit the platelet function (e.g. cyclooxygenase [COX]-1 inhibitors)
* Presence of bleeding diathesis or coagulopathy
* Cumulative anthracycline and anthracenedione exposure as follows: doxorubicin > 450 mg/m^2; epirubicin > 700 mg/m^2; liposomal doxorubicin > 550 mg/m^2; mitoxantrone > 140 mg/m^2
* Proteinuria at baseline; subjects unexpectedly discovered to have >= 1+ proteinuria should undergo a 24-hour urine collection, which must be an adequate collection and must demonstrate =< 500 mg protein/ 24 hours to allow participation in the study
* Cardiac ejection fraction (multigated acquisition scan [MUGA] or echocardiogram) less than the local institution lower limit of normal
* Abnormalities of the cornea based on history (e.g., dry eye syndrome, Sjögren's syndrome), congenital abnormality (e.g., Fuch's dystrophy), abnormal slit-lamp examination using a vital dye (e.g., fluorescein, Bengal-Rose), and/or an abnormal corneal sensitivity test (Schirmer test or similar tear production test)
* Serious, non-healing wound, ulcer, or bone fracture
* Clinically significant cardiovascular disease (e.g., uncontrolled hypertension, myocardial infarction, unstable angina), New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or grade II or greater peripheral vascular disease within 1 year prior to day 0
* Gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, or prior surgical procedures affecting absorption
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with OSI-774
* Human immunodeficiency virus (HIV)-positive patients receiving combination anti-retroviral therapy are excluded from the study
* Patients with recent (within 6 months) arterial thrombotic events, including transient ischemic attack (TIA), cerebrovascular accident (CVA), unstable angina, myocardial infarction (MI), or clinically significant peripheral artery disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2002-12; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maura Dickler, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - UCSF Medical Center-Mount Zion, San Francisco, California
  - Memorial Sloan-Kettering Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Started | 38
Completed | 37
Not Completed | 1
Not completed — Not Treated | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 38

OUTCOME MEASURES:

1. Primary Outcome: Level of EGFR Expression
Description: Estimated at the end of the trial Immunoreactivity will be evaluated qualitatively with regard to intensity as follows: Measured on a scale, ranging from 0-3+ 0=negative (no immunoreactivity)
  1+ - 3+ = positive:
  * faint immunoreactivity (weak staining)
  * intense immunoreactivity (strong staining) Immunohistochemical studies will be performed on the tumor specimen to correlate the anti-tumor efficacy of OSI-774 and bevacizumab with pre-treatment molecular characteristics.
Time Frame: Up to 12 years
Measure: Number; unit: participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 38
participants
  EGFR 0 | 24
  EGFR 1+ | 8
  EGFR 2+ | 4
  EGFR 3+ | 0
  Insufficient tumor tissue | 2

2. Primary Outcome: Response Rate, Defined as Complete Response (CR) + Partial Response (PR), Using the Response Evaluation Criteria in Solid Tumors
Description: Estimated at the end of the trial. Complete Response (CR):Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD 55 Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum LD since the treatment started
Time Frame: Up to 12 years
Measure: Number; unit: participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 37
participants
  Complete Response | 0
  Partial Response | 1
  Stable Disease | 17
  Progression of Disease | 19

3. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).Evaluation of Target Lesions Complete Response (CR):Disappearance of all target lesions Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD
Time Frame: From the time measurement criteria are met for CR and PR until the first date that recurrent or progressive disease is objectively documented, assessed up to 12 years
Measure: Number; unit: months
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 1
months | 52

4. Secondary Outcome: Time to Progression
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From the start of treatment until the first date that recurrent or progressive disease is objectively documented, assessed up to 12 years
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 19
weeks | 11 [8 to 18]

5. Secondary Outcome: Number of Patients Evaluated for Toxicity
Description: graded according to the National Cancer Institute Common Toxicity Criteria version 4.0
Time Frame: up to 12 years
Population: Please see adverse events section.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 38
Participants | 38

6. Secondary Outcome: Participants With Duration of Stable Disease Greater Than or Equal to 6 Months
Description: Duration of stable disease greater than or equal to 6 months
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Number analyzed (Participants) | 17
Participants | 0

7. Other Pre Specified Outcome: HER2 Status
Description: Associations between response and HER2 will be assessed by Fisher's exact test.
Time Frame: Up to 12 years
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Percentage of Cells Staining Positive for EGFR
Description: Associations between markers and tumor response will be assessed by logistic regression analysis. For those markers that are statistically significant, a cut-point analysis will be performed by the maximum chi-square with p-value adjustment method to determine positive values.
Time Frame: Up to 12 years
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Percentage of Cells Staining Positive for Human Epidermal Growth Factor Receptor 3 (HER3)
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Percentage of Cells Staining Positive for Marker of Proliferation Ki-67 (Ki-67)
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Percentage of Cells Staining Positive for p27
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Percentage of Cells Staining Positive for Phosphorylated-mitogen-activated Protein Kinase (MAP) Kinase
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Percentage of Cells Staining Positive for Phosphorylated-v-akt Murine Thymoma Viral Oncogene Homolog 1 (Akt)
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Percentage of Cells Staining Positive for Tumor Protein p53 (p53)
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Percentage of Cells Staining Positive for VEGF
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Percentage of Cells Staining Positive for VEGF Receptor (VEGFR)-1
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Percentage of Cells Staining Positive for VEGFR-2
Description: as for outcome 8
Time Frame: Up to 12 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Treatment (Erlotinib Hydrochloride, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 6/38
Other Adverse Events (participants affected / at risk) | 32/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Erlotinib Hydrochloride, Bevacizumab) (N=38)
General disorders and administration site conditions-other, specify (General disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pain, other (General disorders) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Erlotinib Hydrochloride, Bevacizumab) (N=38)
Alanine aminotransferase increased (Investigations) | 4 (6)
Alkaline phosphatase increased (Investigations) | 5 (6)
Anemia (Blood and lymphatic system disorders) | 3 (12)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Blood bilirubin increased (Investigations) | 8 (10)
Blurred vision (Eye disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Fatigue (General disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypertension (Vascular disorders) | 5 (5)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Infections and infestations - Other, specify (Infections and infestations) | 7 (7)
Lymphocyte count decreased (Investigations) | 7 (19)
Mucositis oral (Gastrointestinal disorders) | 4 (6)
Nail loss (Skin and subcutaneous tissue disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Proteinuria (Renal and urinary disorders) | 3 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 15 (16)
Thromboembolic event (Vascular disorders) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less